CLINICAL TRIAL: NCT00576550
Title: A Randomised Trial of a Moisturising Cream in Preventing Recurrence of Hand Eczema
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ACO Hud Nordic AB (Industry)
Collaborators: Smerud Medical Research International AS (Other)
Responsible Party: Karin Wirén, ACO HUD NORDIC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SMR-1588
Record Dates: First submitted 2007-12-18; First posted 2007-12-19 (Estimated); Last update posted 2008-10-13 (Estimated); Status verified 2007-12

CONDITIONS: Hand Eczema
Keywords: Hand eczema; Prevention
MeSH Terms: interventions — Urea; Betamethasone Valerate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1:1 (Experimental): Part 1 of the study (maintenance part)
  Interventions: Drug: Urea
- 1:2 (No Intervention): Part 1 of the study (maintenance part)
- 2:1 (Experimental): Part 2 of the study (eczema part)
  Interventions: Drug: betamethasone valerate
- 2:2 (Active Comparator): Part 2 of the study (eczema part)
  Interventions: Drug: betamethasone valerate

INTERVENTIONS:
Drug: Urea — Urea cream applied twice daily up to six months
  Other Names: Canoderm 5% kräm
  Arms: 1:1
Drug: betamethasone valerate — Application once daily for two weeks
  Other Names: Betnoderm 0,1 % kräm
  Arms: 2:1
Drug: betamethasone valerate — Application twice daily for two weeks
  Other Names: Betnoderm 0,1 % kräm
  Arms: 2:2

SUMMARY:
The purpose of this study is to investigate whether a moisturizing cream can prevent hand eczema.Patients with previous hand eczema will be studied. In the second part of the study, it will be explored if a treatment regimen of a topical corticosteroid once daily is not inferior to treatment twice daily.

ELIGIBILITY:
Inclusion Criteria:

* Clinically proven history of hand eczema
* At inclusion controlled state of hand eczema (≤3 on Hand Eczema Extent Score, HEES)
* Daily use of moisturising treatment
* Either gender
* Age 18 or above
* Written Informed Consent

Exclusion Criteria:

* Possible allergy to ingredients in the study medications
* At study start active psoriatic lesions or active atopic eczema lesions on the hands. Active bacterial, fungal or viral infection of the hands
* Patients who are pregnant or breast-feeding, or who plan to become pregnant during the course of the study
* Use of any concomitant medication that may interfere with the study related activities or assessment of efficacy
* Any patient related factor suggesting potential poor compliance with study procedures (e.g. psychiatric disorders, history of alcohol or substance abuse)
* Any serious medical condition which, in the opinion of the investigator, may interfere with the evaluation of the results
* Inclusion in a study of an investigational drug within 60 days prior to start of treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2007-10; Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Time to relapse of hand eczema | Up to 6 months

SECONDARY OUTCOMES:
The number of patients showing clearance of hand eczema after betamethasone treatment once versus twice daily | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gro Moerk, MD, Principal Investigator — Rikshospitalet, Oslo
Locations (3):
- Norway (3):
  - Medi 3 Innlandet, Hamar
  - Colosseumklinikken, Oslo
  - Dr Funks hudklinikk, Oslo